CLINICAL TRIAL: NCT05504577
Title: Blood-saving Effect of Kaolin-based Hemostatic Gauze Combined With Intravenous Tranexamic Acid in Total Knee Arthroplasty
Brief Title: Kaolin-based Hemostatic Gauze in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMRPG8M0261
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Total Blood Loss; Arthropathy of Knee Joint
Keywords: Postoperative blood loss; Total knee arthroplasty; kaolin-impregnated gauze; tranexamic acid
MeSH Terms: conditions — Exsanguination; Postoperative Hemorrhage | interventions — Tranexamic Acid; Tranylcypromine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- QCG group (Experimental): After the prosthesis are all implanted, apply the QCG (Quikclot Z-fold hemostatic gauze, Z-Medica, Wallingford, CT, USA) into the joint space. Compress the knee joint by elastic bandage. Deflate the tourniquet for 10 minutes, then remove the QCG from the knee joint and throughout check bleeders before closure of the joint capsule. Tranexamic acid 1g is intravenously injected at 10 mins before tourniquet deflation
  Interventions: Drug: Tranexamic acid injection; Device: apply the QCG
- Surgical gauze group (Active Comparator): After the prosthesis are all implanted, apply the surgical gauze into the joint space. Compress the knee joint by elastic bandage. Deflate the tourniquet for 10 minutes, then remove the gauze from the joint and throughout check bleeders before closure of the joint capsule. Tranexamic acid 1g is intravenously injected at 10 mins before tourniquet deflation
  Interventions: Drug: Tranexamic acid injection; Device: apply surgical gauze
- Control group (Placebo Comparator): fter the prosthesis are all implanted, we close the joint capsule directly. Tranexamic acid 1g is intravenously injected at 10 mins before tourniquet deflation. .
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — Tranexamic acid 1g is intravenously injected at 10 mins before tourniquet deflation. .
  Other Names: transamine injection
Device: apply the QCG — apply the QCG (Quikclot Z-fold hemostatic gauze, Z-Medica, Wallingford, CT, USA) into the joint space. Compress the knee joint by elastic bandage. Compress the knee joint by elastic bandage. Deflate the tourniquet for 10 minutes
  Arms: QCG group
Device: apply surgical gauze — apply the normal surgical gauze into the joint space. Compress the knee joint by elastic bandage. Deflate the tourniquet for 10 minutes
  Arms: Surgical gauze group

SUMMARY:
This study is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of combination of intravenous TXA and QCG in a primary TKA procedure.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is associated with considerable blood loss and increasing needs for allogenic blood transfusion. Previous studies demonstrated a transfusion rates ranging from 10% to 38% after standard TKAs. Tranexamic acid (TXA), an inhibitor of fibrinolysis, was reportedly effective reducing blood loss after standard TKA. Our previous experiences in minimally invasive (MIS) TKA showed that intraoperative intravenous infusion of TXA reduced 45% of postoperative blood loss and needs for transfusion from 20% to 4%. Our study demonstrated that an equal efficacy of intraarticular topical TXA in blood conservation compared with intravenous infusion of TXA.

In addition to TXA, the Quikclot sponge (QCG; Z-Medica, Wallingford, CT, USA) is a newly developed hemostatic agent employing an inorganic mineral (kaolin). The QCG has predominantly been used in combat settings and trauma surgery. Recently, the application of QCG in interventional procedures, and non-orthopedic surgeries was reported. Literature describing the use of QCG as an alternative approach to achieve hemostasis in the field of orthopedics is limited. There is no study to investigate the blood-saving effect of QCG in a TKA procedure, especially in combined with TKA. Therefore we conduct the study to understand the efficacy of this sponge on blood conservation in TKA We believe that combination with the two different mechanism of blood-conservation agents can bring a synergistic effect in blood saving after TKA. Our purpose of this study therefore is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of QCG combined with TXA use.

Material and Methods:

The patients who are enrolled in this study will be randomly assigned into three groups. We plan to recruit 60 patients in each group (total case number is 120). The first group will be treated by application of QCG in joint space and TXA 1g intravenous injection before tourniquet deflation. The second group will be treated by application of normal gauze in joint space and TXA 1g intravenous injection before tourniquet deflation. The third group will be treated only TXA 1g intravenously injection alone before tourniquet deflation. We will observe whether there is difference in the blood-conservation effect by total blood loss calculation, hemoglobin loss and transfusion requirement between these three groups. Besides, any complications including VTE, deep infection, wound complications within postoperative 3 months will be recorded.

Study years: two years

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced osteoarthritis of the knee and undergo primary unilateral minimally invasive TKA
* Age > 50 years and < 90 years
* Failure of medical treatment or rehabilitation
* Hemoglobin ≧ 11g/dl
* No use of non-steroid anti-inflammatory agent, antiplatelets or anticoagulants at least 3 days before operation

Exclusion Criteria:

1. Preoperative Hemoglobin <11 g/dl
2. History of infection or intraarticular fracture of the affective knee
3. Renal function deficiency (GFR <30 ml/min/1.73m2)
4. Elevated liver enzyme (AST/ALT level are more than twice normal range) , history of liver cirrhosis, impaired liver function(elevated total bilirubin level) and coagulopathy (including long-term use anticoagulant)
5. History of deep vein thrombosis, ischemic heart disease or stroke, in which life-long oral anticoagulant are required.
6. Contraindications of tranexamic acid, or rivaroxaban
7. Allergy to tranexamic acid, kaolin, rivaroxaban, or the excipients
8. History of heparin-induced thrombocytopenia (HIT)
9. Coagulopathy or bleeding tendency caused by organ dysfunction, such as cirrhosis, bone marrow suppression etc.
10. Patient who have active bleeding disorder, such as intracranial hemorrhage, upper GI bleeding, hematuria..

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Total Blood Loss | Preoperative day to postoperative day 4
  The total blood loss was calculated according to Nadler et al, which uses maximum postoperative decrease of the Hb level adjusted for weight and height of the patient. Total blood loss consists of amount of blood loss calculated from the maximum Hb loss and amount of blood transfused

SECONDARY OUTCOMES:
Blood transfusion rate | To three months after operation
  We will record the event of blood transfusion, and calculate the incidence of transfusion
All symptomatic thrombotic events including deep vein thrombosis, pulmonary embolism | To three months after operation
  We will record all symptomatic thrombotic events including deep vein thrombosis, pulmonary embolism in our study, and calculate the incidence of them

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Wen Wang, MD, Study Director — Department of Orthopaedic Surgery, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bong MR, Patel V, Chang E, Issack PS, Hebert R, Di Cesare PE. Risks associated with blood transfusion after total knee arthroplasty. J Arthroplasty. 2004 Apr;19(3):281-7. doi: 10.1016/j.arth.2003.10.013. PMID 15067638
- [Background] Bierbaum BE, Callaghan JJ, Galante JO, Rubash HE, Tooms RE, Welch RB. An analysis of blood management in patients having a total hip or knee arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):2-10. doi: 10.2106/00004623-199901000-00002. PMID 9973048
- [Background] Goodnough LT, Verbrugge D, Marcus RE. The relationship between hematocrit, blood lost, and blood transfused in total knee replacement. Implications for postoperative blood salvage and reinfusion. Am J Knee Surg. 1995 Summer;8(3):83-7. PMID 7552610
- [Background] Tanaka N, Sakahashi H, Sato E, Hirose K, Ishima T, Ishii S. Timing of the administration of tranexamic acid for maximum reduction in blood loss in arthroplasty of the knee. J Bone Joint Surg Br. 2001 Jul;83(5):702-5. doi: 10.1302/0301-620x.83b5.11745. PMID 11476309
- [Background] Alvarez JC, Santiveri FX, Ramos I, Vela E, Puig L, Escolano F. Tranexamic acid reduces blood transfusion in total knee arthroplasty even when a blood conservation program is applied. Transfusion. 2008 Mar;48(3):519-25. doi: 10.1111/j.1537-2995.2007.01564.x. Epub 2007 Dec 7. PMID 18067499
- [Background] Petaja J, Myllynen P, Myllyla G, Vahtera E. Fibrinolysis after application of a pneumatic tourniquet. Acta Chir Scand. 1987 Nov-Dec;153(11-12):647-51. PMID 3124428
- [Background] Kambayashi J, Sakon M, Yokota M, Shiba E, Kawasaki T, Mori T. Activation of coagulation and fibrinolysis during surgery, analyzed by molecular markers. Thromb Res. 1990 Oct 15;60(2):157-67. doi: 10.1016/0049-3848(90)90294-m. PMID 2149215
- [Background] Hiippala S, Strid L, Wennerstrand M, Arvela V, Mantyla S, Ylinen J, Niemela H. Tranexamic acid (Cyklokapron) reduces perioperative blood loss associated with total knee arthroplasty. Br J Anaesth. 1995 May;74(5):534-7. doi: 10.1093/bja/74.5.534. PMID 7772427
- [Background] Benoni G, Fredin H. Fibrinolytic inhibition with tranexamic acid reduces blood loss and blood transfusion after knee arthroplasty: a prospective, randomised, double-blind study of 86 patients. J Bone Joint Surg Br. 1996 May;78(3):434-40. PMID 8636182
- [Background] Lin PC, Hsu CH, Chen WS, Wang JW. Does tranexamic acid save blood in minimally invasive total knee arthroplasty? Clin Orthop Relat Res. 2011 Jul;469(7):1995-2002. doi: 10.1007/s11999-011-1789-y. Epub 2011 Feb 1. PMID 21286886
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on blood loss and transfusion rate in primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1080-3. doi: 10.1016/j.arth.2012.11.016. Epub 2013 Mar 28. PMID 23541868
- [Background] Chimento GF, Huff T, Ochsner JL Jr, Meyer M, Brandner L, Babin S. An evaluation of the use of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):74-7. doi: 10.1016/j.arth.2013.06.037. PMID 24034510
- [Background] Konig G, Hamlin BR, Waters JH. Topical tranexamic acid reduces blood loss and transfusion rates in total hip and total knee arthroplasty. J Arthroplasty. 2013 Oct;28(9):1473-6. doi: 10.1016/j.arth.2013.06.011. Epub 2013 Jul 23. PMID 23886406
- [Background] Georgiadis AG, Muh SJ, Silverton CD, Weir RM, Laker MW. A prospective double-blind placebo controlled trial of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):78-82. doi: 10.1016/j.arth.2013.03.038. Epub 2013 Jul 29. PMID 23906869
- [Background] Yen SH, Lin PC, Chen B, Huang CC, Wang JW. Topical Tranexamic Acid Reduces Blood Loss in Minimally Invasive Total Knee Arthroplasty Receiving Rivaroxaban. Biomed Res Int. 2017;2017:9105645. doi: 10.1155/2017/9105645. Epub 2017 Dec 19. PMID 29410968
- [Background] Rajagopalan V, Chouhan RS, Pandia MP, Lamsal R, Rath GP. Effect of Intraoperative Blood Loss on Perioperative Complications and Neurological Outcome in Adult Patients Undergoing Elective Brain Tumor Surgery. J Neurosci Rural Pract. 2019 Oct;10(4):631-640. doi: 10.1055/s-0039-3399487. Epub 2019 Dec 11. PMID 31831982
- [Background] Walsh PN. The effects of collagen and kaolin on the intrinsic coagulant activity of platelets. Evidence for an alternative pathway in intrinsic coagulation not requiring factor XII. Br J Haematol. 1972 Apr;22(4):393-405. doi: 10.1111/j.1365-2141.1972.tb05687.x. No abstract available. PMID 5028124
- [Background] Gegel BT, Austin PN, Johnson AD. An evidence-based review of the use of a combat gauze (QuikClot) for hemorrhage control. AANA J. 2013 Dec;81(6):453-8. PMID 24597007
- [Background] Motamedi MH, Sagafinia M. QuickClot combat gauze use for hemorrhage control in military trauma. Prehosp Disaster Med. 2011 Jun;26(3):237. doi: 10.1017/S1049023X11006273. No abstract available. PMID 22107778
- [Background] Travers S, Lefort H, Ramdani E, Lemoine S, Jost D, Bignand M, Tourtier JP. Hemostatic dressings in civil prehospital practice: 30 uses of QuikClot Combat Gauze. Eur J Emerg Med. 2016 Oct;23(5):391-4. doi: 10.1097/MEJ.0000000000000318. PMID 26351975
- [Background] Shina A, Lipsky AM, Nadler R, Levi M, Benov A, Ran Y, Yitzhak A, Glassberg E. Prehospital use of hemostatic dressings by the Israel Defense Forces Medical Corps: A case series of 122 patients. J Trauma Acute Care Surg. 2015 Oct;79(4 Suppl 2):S204-9. doi: 10.1097/TA.0000000000000720. PMID 26406432
- [Background] Trabattoni D, Gatto P, Bartorelli AL. A new kaolin-based hemostatic bandage use after coronary diagnostic and interventional procedures. Int J Cardiol. 2012 Apr 5;156(1):53-4. doi: 10.1016/j.ijcard.2010.10.030. Epub 2010 Nov 18. PMID 21087799
- [Background] Derkay CS, Baydoun HA, Stone L. Intraoperative Use of QuikClot During Adenotonsillectomy: A Prospective Pediatric Trial. Ann Otol Rhinol Laryngol. 2015 May;124(5):384-91. doi: 10.1177/0003489414560432. Epub 2014 Nov 25. PMID 25423961
- [Background] Patel SA, Martin M, Chamales I. Vaginal hemorrhage from transobturator sling controlled with QuikClot combat gauze. Mil Med. 2012 Aug;177(8):997-8. doi: 10.7205/milmed-d-11-00429. PMID 22934384
- [Background] Schmid BC, Rezniczek GA, Rolf N, Maul H. Postpartum hemorrhage: use of hemostatic combat gauze. Am J Obstet Gynecol. 2012 Jan;206(1):e12-3. doi: 10.1016/j.ajog.2011.09.018. Epub 2011 Sep 24. PMID 22011588
- [Background] Abbott EM, Nandyala SV, Schwend RM. Does a kaolin-impregnated hemostatic dressing reduce intraoperative blood loss and blood transfusions in pediatric spinal deformity surgery? Spine (Phila Pa 1976). 2014 Sep 1;39(19):E1174-80. doi: 10.1097/BRS.0000000000000466. PMID 24921838
- [Background] Kim K, Shim H, Jung PY, Kim S, Choi YU, Bae KS, Lee JK, Jang JY. Effectiveness of kaolin-impregnated hemostatic gauze use in preperitoneal pelvic packing for patients with pelvic fractures and hemodynamic instability: A propensity score matching analysis. PLoS One. 2020 Jul 24;15(7):e0236645. doi: 10.1371/journal.pone.0236645. eCollection 2020. PMID 32706824